CLINICAL TRIAL: NCT02125253
Title: A Blinded, Randomized, Placebo-Controlled, Parallel Group, Multi-Site Study to Compare the Therapeutic Equivalence of Mometasone Furoate Nasal Spray, 50 mcg (Amneal Pharmaceuticals LLC) With NASONEX® Nasal Spray (Schering Corporation) in the Relief of the Signs and Symptoms of Seasonal Allergic Rhinitis
Brief Title: Study to Compare the Therapeutic Equivalence of Mometasone Furoate Nasal Spray, 50 mcg With Nasonex Nasal Spray in the Relief of the Signs and Symptoms of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amneal Pharmaceuticals, LLC (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AM-MMS-001
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mometasone Furoate Nasal Spray, 50 mcg (Experimental): Mometasone Furoate Nasal Spray, 50 mcg. 4 actuations per day for 14 days.
  Interventions: Drug: Mometasone Furoate Nasal Spray, 50 mcg
- Nasonex Nasal Spray, 50 mcg (Active Comparator): Nasonex (mometasone furoate monohydrate) Nasal Spray, 50 mcg. 4 actuations per day for 14 days.
  Interventions: Drug: Nasonex Nasal Spray, 50 mcg
- Placebo Nasal Spray (Placebo Comparator): Placebo of Mometasone Furoate Nasal Spray. 4 actuations per day for 14 days.
  Interventions: Drug: Placebo Nasal Spray

INTERVENTIONS:
Drug: Mometasone Furoate Nasal Spray, 50 mcg — a metered-dose, manual pump spray unit containing an aqueous suspension of mometasone furoate
  Arms: Mometasone Furoate Nasal Spray, 50 mcg
Drug: Nasonex Nasal Spray, 50 mcg — a metered-dose, manual pump spray unit containing an aqueous suspension of mometasone furoate monohydrate
  Arms: Nasonex Nasal Spray, 50 mcg
Drug: Placebo Nasal Spray — a metered-dose, manual pump spray unit containing an aqueous suspension
  Arms: Placebo Nasal Spray

SUMMARY:
To evaluate the therapeutic equivalence of the lest formulation of Mometasone Furoate Nasal Spray, 50 mcg to the marketed formulation NASONEX® (mometasone furoate monohydrate) Nasal Spray, 50 mcg/actuation in patients with seasonal allergic rhinitis

ELIGIBILITY:
Inclusion Criteria:

* If female and of child-bearing potential, have a negative urine pregnancy test and is prepared to abstain from sexual intercourse or use a reliable method of contraception during the study
* Documented positive allergic skin test, performed within the previous 12 months, to one or more of the allergens in season at the time the study is being conducted.
* A minimum of two consecutive years of previous history of seasonal allergic rhinitis to the pollen/allergen in season at the time the study is being conducted.
* A score of at least 6 on the reflective Total Nasal Symptom Score (rTNSS) and a minimum score of at least 2 for "nasal congestion" and a minimum score of at least 2 for one of the remaining 3 symptoms representing the 12hours prior to the screening visit.
* An average composite score of at least 6 on the rTNSS and a minimum score of at least 2 for "nasal congestion" and a minimum score of at least 2 for one of the remaining 3 symptoms representing the last 3 days of the 7-day placebo lead-in period before the randomization visit and the morning of the first day.

of the randomization visit.

Exclusion Criteria:

* Females who are pregnant, lactating or likely to become pregnant during the study.
* Negative or lack of documented skin allergen test (performed within the previous 12 months) to at least one of the allergens in season at the time the study is being conducted.
* Patients who suffer from chronic signs and symptoms of Perennial Allergic Rhinitis, unless the investigator assesses that the patient's current signs and symptoms are a clear exacerbation of Seasonal Allergic Rhinitis (SAR) rather than chronic PAR.
* Patients who suffer only from perennial allergic rhinitis or seasonal allergic rhinitis to a different allergen than that in season at the time the study is conducted.
* Previous history of less than 2 years of seasonal allergic rhinitis to the pollen/allergen in season at the time the study is being conducted.
* Any patient who meets the minimum rTNSS requirements at the start of the placebo lead-in period but no longer meets the requirements prior to the randomized active treatment period of the study cannot continue in the active treatment period.
* History of asthma over the previous two years that required chronic therapy. Occasional acute or mild exercise induced asthma will be allowable on the condition that the treatment of the attacks is restricted to beta-agonists only.
* Patients with nasal conditions, including infectious rhinitis, rhinitis medicamentosa or atrophic rhinitis.
* Clinically significant nasal deformity or any recent nasal surgery or trauma that has not completely healed.
* Sinus infection within the previous 30 days or history of reoccurring sinus infections.
* Patient has started immunotherapy or changed their dose of immunotherapy within 30 days of the first placebo lead-in dose or is likely to have to start immunotherapy, or change their current dose during the study.
* Treatment for oral Candidiasis within 30 days of starting the study or a current oral Candidiasis infection.
* Upper respiratory tract infection within the previous 30 days.
* Patients with a history of tuberculosis.
* Patients with the presence of glaucoma, cataracts, ocular herpes simplex, conjunctivitis or other eye infection not related to the diagnosis of SAR within 14 days of enrollment.
* The patient has had recent exposure (30 days) or was at risk of being exposed to chicken pox or measles.
* Patients with any untreated fungal, bacterial, systemic viral infections within the previous 30 days.
* Use of any ophthalmic steroids within 14 days or nasal, inhaled or systemic steroids within 30 days of the study start.
* Use of the reference product, Nasonex® within 3 months of the study start.
* Use of intranasal or systemic second-generation anti-histamines within10 days of enrollment.
* Use of intranasal cromolyn within 14 days of enrollment.
* Use of intranasal or systemic first-generation anti-histamines, leukotriene receptor antagonists or other nasal decongestants within 3 days of enrollment.
* Use of any tricyclic anti-depressant within 30 days of enrollment
* Patients with attention-deficit disorder being treated with methylphenidate containing products that have not been on a stable dosing regimen for at least the 30 previous days and who cannot remain on the same dosing regimen throughout the study.
* Desensitization therapy to the seasonal allergen that is causing the patients allergic rhinitis within the previous 6 months.
* Previous SAR and/or PAR that has proven unresponsive to steroid therapy.
* Any known hypersensitivity to mometasone, other steroids or any of the components of the study nasal spray.
* Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participating or could jeopardize the integrity of the study evaluations.
* Receipt of any drug as part of a research study within 30 days prior to the first placebo lead-in dose.
* Planned travel outside of the local area for more than 2 consecutive days or 3 days in total, during the patient's participation in the study.
* Previous participation in this study.
* The patient currently smokes cigarettes, cigars, and/or pipes and is a heavy smoker
* The patient shares a household with another patient currently enrolled in this study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 811 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline rTNSS | Days 1 - 14
  Change from baseline in average AM/PM reflective Total Nasal Symptom Score (rTNSS) over Days 1 to 14
Total Nasal Symptom Score (TNSS) | Days 1 - 14
  The sum of patient-rated severity scores for four allergy symptoms : runny nose, nasal congestion, itchy nose, and sneezing based on a 4-point scale.

SECONDARY OUTCOMES:
Change in Baseline iTNSS | Days 1 - 14
  Change from baseline in average instantaneous Total Nasal Symptom Score (iTNSS) over Days 1 to 14.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Gallicano, PhD, Study Chair — Novum Pharmaceutical Reserach Services
Locations (10):
- United States (10):
  - Isis Clinical Research, Austin, Texas
  - Austin Clinical Research, Austin, Texas
  - Sirius Clinical Research, Austin, Texas
  - Kerrville Research Associates, Kerrville, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Allergy & Asthma Research Center, San Antonio, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Sylvania Research, San Antonio, Texas
  - Allergy & Asthma Care of Waco, Waco, Texas